CLINICAL TRIAL: NCT04708769
Title: Evaluating the EVO Treatment Optimized for Resource Constraints: Elements Vital to Treat Obesity.
Brief Title: Elements Vital to Treat Obesity Study
Acronym: EVO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Angela Fidler Pfammatter, PhD, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00212742
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: Weight Loss; Diet; Physical Activity; Self Monitoring; Mobile Health
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smartphone App Participants (APP) (Experimental): Smartphone application, diet and activity goals, online lessons, brief remote sessions with a Health Promotionist
  Interventions: Behavioral: Smartphone App Participants (APP)
- Diabetes Prevention Program Participants (DPP) (Experimental): Participant program manual, diet and activity logs, hour long remote sessions with a Health Promotionist
  Interventions: Behavioral: Diabetes Prevention Program Participants (DPP)

INTERVENTIONS:
Behavioral: Smartphone App Participants (APP) — Participants will receive calorie, fat, and physical activity goals, a Smartphone application for self-monitoring their diet, activity and weight, online educational readings, and brief bi-weekly remote health sessions with a Health Promotionist. They will also be provided with a wireless bluetooth scale and portable blood pressure machine.
  Arms: Smartphone App Participants (APP)
Behavioral: Diabetes Prevention Program Participants (DPP) — In accordance with the Center for Disease Control curriculum, participants will receive a participant log for tracking physical activity, food intake, and weight, a paper participant guide with worksheets, logs, and psycho-educational materials, and 16 hour long remote sessions with a Health Promotionist. They will also be provided with a wireless bluetooth scale and portable blood pressure machine.
  Arms: Diabetes Prevention Program Participants (DPP)

SUMMARY:
The overall objective of this study is to evaluate the first rigorously optimized, remotely delivered treatment for obesity against the current gold standard treatment in a head-to-head randomized controlled trial. The investigators will be comparing the previously developed and optimized behavioral weight loss intervention (APP) to the Diabetes Prevention Program (DPP), to evaluate program weight-loss success and cost-effectiveness.

DETAILED DESCRIPTION:
The proposed study seeks to determine if the APP program is an effective, resource-sensitive strategy to manage weight for obesity, as compared to the DPP program. During the 24-week active intervention phase, participants will be randomized to one of two treatments: 1) APP, wherein participants receive calorie, fat, and physical activity goals via a Smartphone application for self-monitoring, online educational readings, and biweekly sessions with a Health Promotionist; or 2) DPP, wherein participants are guided to self-monitor their physical activity, food intake, and weight via a participant log, and are guided through 16 sessions by a Health Promotionist. Assessments to track progress will occur remotely at the 3-month, 6-month, and 12-month time points of the program.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-45
* Weight stable
* Own a Smartphone and be willing to install our Smartphone app
* Willing to conduct video conference calls with study staff

Exclusion Criteria:

* Enrolled in any formal weight loss program
* Taking anti-obesity medications
* Not taking medications that may cause weight gain
* Unstable medical conditions
* Diabetes requiring insulin supplementation
* Crohn's Disease
* Diagnosis of obstructive sleep apnea requiring intervention (i.e., CPAP)
* Assistive devices for mobility
* Hospitalizations for a psychiatric disorder within the past 5 years
* Cardiovascular disease symptoms while performing moderate intensity exercise
* Pregnancy, trying to get pregnant, or lactating.
* Bulimia or binge eating disorder
* Reports of active suicidal ideation
* Current substance abuse or dependence besides nicotine dependence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight | Baseline to 6-Months
  Participant change in weight, in kilograms, from baseline to 6-months.

SECONDARY OUTCOMES:
Costs of treatment | 12 Months
  Costs of EVO versus DPP implementation

CONTACTS AND LOCATIONS:
Overall Officials: Angela Pfammatter, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882